CLINICAL TRIAL: NCT02302261
Title: Using Pleth Variability to Triage Asthmatics in the Pediatric ED
Brief Title: Pleth Variability and Asthma Severity in Children
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Ariel Brandwein, Pediatric Critical Care Fellow, Northwell Health
Other Study IDs: 14-572
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Status Asthmaticus
Keywords: Pulsus paradoxus
MeSH Terms: conditions — Status Asthmaticus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Status Asthmaticus: Any patient presenting to the ED with status asthmaticus.

SUMMARY:
Research has shown that pleth variability can be used to assess asthma severity in children with status asthmaticus. The investigators would like to use an FDA-cleared monitor (Masimo Radical 7) which measures Pleth Variability Index (PVI) to see if the degree of PVI can be used to help triage patients who present to the pediatric ED in status asthmaticus.

DETAILED DESCRIPTION:
Patients with asthma have obstruction to exhalation resulting in hyperinflation of their lungs. This hyperinflation results in a phenomenon known as pulsus paradoxus in which the physiologic drop in blood pressure normally seen with inhalation is exaggerated. Studies have shown that patients with more severe asthma exacerbations (i.e. more hyperinflation) have a greater degree of pulsus paradoxus. Typically, pulsus paradoxus is measured using a sphygmomanometer, however, researchers have demonstrated that it can also accurately be measured using plethysmography, a term known as pleth variability index (PVI). Using this concept, Arnold et al (2008, 2010) showed that a greater degree of pulsus paradoxus correlates with asthma severity.

The investigators' study aims to simplify the association between PVI and asthma severity. The investigators hypothesize the following:

1. Patients with a higher admission PVI will have a higher likelihood of being admitted to the hospital.
2. Patients admitted to the Intensive Care Unit (PICU) will have a higher PVI than patients admitted to a floor.
3. PVI can be accurately used to gauge response to bronchodilator/anti-inflammatory therapy.
4. PVI is as effective as respiratory severity score in predicting asthma severity and in gauging response to bronchodilator therapy.

To do this the investigators will recruit children who present to the pediatric ED in status asthmaticus. They will be connected to a Masimo Radical 7 monitor upon admission to the ED and then again 4 hours later. In addition the investigators will calculate respiratory severity scores at those same time intervals. The investigators will then look at the disposition of the patient upon leaving the ED: discharge to home, admission to an inpatient floor or admission to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma or reactive airway disease upon leaving the ED
* Greater than 10 kg

Exclusion Criteria:

* Patients in whom effective pulse oximetry tracings cannot be obtained
* Patients who are diagnosed with conditions other than asthma/reactive airway disease that are known to cause pulsus paradoxus

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will study patients who present to the pediatric ED at Cohen Children's Medical Center of NY with status asthmaticus.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Disposition from ED | 4 hours
  Determine whether a patient was discharged from the ED, admitted to an inpatient floor or admitted to the ICU.

SECONDARY OUTCOMES:
Comparison to respiratory severity score | 4 hours
  Is PVI as effective as RSS in determining asthma severity
Change in disposition within 24 hours | 1 week
  Determine if a patient who was discharged home from the ED required readmission to the ED within 1 week. Determine if a patient admitted to the floor or ICU required a change in level of care in the first 24 hours of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Brandwein, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center of NY, New Hyde Park, New York, United States

REFERENCES:
- [Background] Arnold DH, Gebretsadik T, Minton PA, Higgins S, Hartert TV. Assessment of severity measures for acute asthma outcomes: a first step in developing an asthma clinical prediction rule. Am J Emerg Med. 2008 May;26(4):473-9. doi: 10.1016/j.ajem.2007.05.026. PMID 18410819
- [Background] Arnold DH, Jenkins CA, Hartert TV. Noninvasive assessment of asthma severity using pulse oximeter plethysmograph estimate of pulsus paradoxus physiology. BMC Pulm Med. 2010 Mar 29;10:17. doi: 10.1186/1471-2466-10-17. PMID 20350320
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Clark JA, Lieh-Lai M, Thomas R, Raghavan K, Sarnaik AP. Comparison of traditional and plethysmographic methods for measuring pulsus paradoxus. Arch Pediatr Adolesc Med. 2004 Jan;158(1):48-51. doi: 10.1001/archpedi.158.1.48. PMID 14706958
- [Background] Frey B, Freezer N. Diagnostic value and pathophysiologic basis of pulsus paradoxus in infants and children with respiratory disease. Pediatr Pulmonol. 2001 Feb;31(2):138-43. doi: 10.1002/1099-0496(200102)31:23.0.co;2-r. PMID 11180690
- [Background] Rayner J, Trespalacios F, Machan J, Potluri V, Brown G, Quattrucci LM, Jay GD. Continuous noninvasive measurement of pulsus paradoxus complements medical decision making in assessment of acute asthma severity. Chest. 2006 Sep;130(3):754-65. doi: 10.1378/chest.130.3.754. PMID 16963672